CLINICAL TRIAL: NCT00669578
Title: A Phase I/II, Prospective, Open-Label Study to Determine the Safety and Efficacy of CC-4047 in Patients With Primary, Post Polycythemia Vera, or Post Essential Thrombocythemia Myelofibrosis®
Brief Title: CC-4047 in Treating Patients With Myelofibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC078B; P30CA015083 (NIH); MC078B (Other: Mayo Clinic Cancer Center); NCI-2009-01331 (Registry Identifier: NCI-CTRP); 07-005317 (Other: Mayo Clinic IRB); PO-MMM-PI-0007 (Other: Celgene Protocol)
Record Dates: First submitted 2008-04-29; First posted 2008-04-30 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Chronic Myeloproliferative Disorders; Secondary Myelofibrosis
Keywords: secondary myelofibrosis; polycythemia vera; essential thrombocythemia; primary myelofibrosis
MeSH Terms: conditions — Myeloproliferative Disorders; Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CC-4047 (Experimental)
  Interventions: Drug: CC-4047

INTERVENTIONS:
Drug: CC-4047 — CC-4047: taken orally each day in a 28 day cycle.

SUMMARY:
RATIONALE: Biological therapies, such as CC-4047, may stimulate the immune system in different ways and stop cancer cells from growing. CC-4047 may also stop the growth of cancer cells by blocking blood flow to the cancer.

PURPOSE: This trial is studying the side effects and best dose of CC-4047 and to see how well it works in treating patients with myelofibrosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Phase I:

Primary

* To determine the Maximum Tolerated Dose of CC-4047 in the treatment of Primary, Post Polycythemia Vera, or Post Essential Thrombocythemia Myelofibrosis (PMF, post-PV MF, or post-ET MF).

Phase II:

Primary

* Best overall response as determined by International Working Group Criteria over the first 6 cycles (168 days) of study treatment.

Secondary

* Safety (type, frequency, severity [National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0] of adverse events (AEs), and relationship of AEs to CC-4047.
* Duration of response.
* Time to response.
* Best overall response as determined by International Working Group Criteria over the first 12 cycles (336 days) of study treatment.

OUTLINE: Patients receive oral CC-4047. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 28 days and then every 6 months for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary and post essential thrombocythemia (ET) or post polycythemia vera (PV) myelofibrosis requiring therapy

  * De novo presentation (i.e., agnogenic myeloid metaplasia AND post ET or post PV myelofibrosis)
  * Developed after an antecedent history of PV (i.e., post polycythemic myeloid metaplasia) or essential polycythemia (i.e., post thrombocythemic myeloid metaplasia)
* Total hemoglobin < 10 g/dL OR transfusion dependent anemia (defined by a history of ≥ 2 units of red blood cell (RBC) transfusions within the past 28 days for hemoglobin < 8.5 g/dL that was not associated with overt bleeding) OR marked splenomegaly (e.g., ≥ 10 cm below costal margin)

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) ≥ 500/μL
* Platelet count ≥ 20,000/μL
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3 times upper limit of normal (ULN) (≤ 5 times ULN if attributed to hepatic extramedullary hematopoiesis)
* Total bilirubin ≤ 3 times ULN OR direct bilirubin ≤ 2 times ULN
* Serum creatinine ≤ 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception for ≥ 28 days before, during, and for ≥ 28 days after completion of study treatment
* Agrees to abstain from donating blood, semen, or sperm during and for ≥ 28 days after completion of study treatment
* Willing to undergo transfusion of blood products (if applicable)
* Able to complete questionnaire(s) alone or with assistance
* No known HIV positivity, hepatitis B carrier, or active hepatitis C infection
* No serious medical condition, psychiatric illness, or any other condition, including the presence of laboratory abnormalities, that (as judged by the treating physician) would preclude giving informed consent or participating in the study or confound the ability to interpret data from the study
* No other active malignancies, except basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast
* No active deep vein thrombosis or pulmonary embolism that has not been therapeutically anticoagulated

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* No prior CC-4047
* More than 28 days since prior growth factors, cytotoxic chemotherapeutic agents (e.g., hydroxyurea or anagrelide), corticosteroids, or experimental drugs or therapies
* No other concurrent experimental drugs or therapies or cytotoxic chemotherapeutic agents (e.g., hydroxyurea or anagrelide) for myelofibrosis
* No concurrent growth factors (including erythropoietin) for myelofibrosis, except G-CSF or pegfilgrastim
* No concurrent chronic use (i.e., > 2 weeks) of more than physiologic doses of corticosteroids (dose equivalent to > 10 mg/day of prednisone)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2010-07-07 (Actual); Study Completion 2019-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben A. Mesa, MD, Principal Investigator — Mayo Clinic; Ayalew Tefferi, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened June 2008 and accrued 12 Phase I participants and 65 Phase II participants before being closed in January 2010.
Pre-assignment Details: Participants were accrued to the Phase I portion of this study in each of the 2.5, 3.0, and 3.5 mg dose cohorts. Dose Limiting Toxicities (DLT) were observed at the 3.5 mg level, and the 3 mg level was confirmed as the maximum tolerated dose. However, efficacy was not improved at higher doses and the most effective dose level was deemed 0.5 mg/day.
Groups:
- Phase I: Participants were accrued to the Phase I portion of this study in each of the 2.5, 3.0, and 3.5 mg dose cohorts to determine the Maximum Tolerated Dose (MTD). Dose limiting Toxicities (DLT) were observed at the 3.5 mg level, and the 3 mg level was confirmed as the maximum tolerated dose. For this study a DLT was defined as a grade 4 hematologic toxicity, a grade 3 or higher febrile neutropenia, or a grade 3 or higher non-hematologic toxicity.
- Phase II: All patients enrolled to this phase II arm started treatment at 0.5mg/day with CC-4047 every day of each 28 day cycle.
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 12 | 65
Completed | 12 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase II | Phase I | Total
Number analyzed (Participants) | 65 | 12 | 77
Age, Continuous [Median (Full Range); unit: years] | 68 (9.7) [42 to 87] | 66 [51 to 83] | 67 [42 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 7 | 25
  Male | 47 | 5 | 52
Region of Enrollment [Number; unit: participants]
  United States | 65 | 12 | 77

OUTCOME MEASURES:

1. Primary Outcome: Determine the Maximum Tolerated Dose of CC-4047
Description: Starting at a dose level of 2.5 mg/d on days 1-21 in every 28 day cycle, participants were accrued in cohorts of three to assess dose limiting toxicities (DLT) and determine the maximum tolerated dose (MTD). Dose escalation at increments of 0.5 mg/d was done if no subject had a DLT (a grade 4 or higher hematologic toxicity or a grade 3 or higher febrile neutropenia or a grade 3 or higher non-hematologic toxicity) in cycle 1. Subsequent cohorts were treated until the maximum tolerated dose (MTD) was reached (dose level before that which results in a DLT in >1 of 6 subjects). Subsequent participants were treated at the MTD, those without response at the MTD after 3 cycles were lowered to the minimal efficacious dose (MED) of 0.5 mg daily. Here, we are reporting the percentage of participants in Phase I with a DLT at each dose level.
Time Frame: The first 28-day cycle of treatment.
Population: None of the Phase II participants were evaluable for this endpoint. For the Phase I portion of this study, three participants were accrued at a 2.5 mg/day dose level, six at the 3.0 mg/day dose level, and three at the 3.5 mg/day dose level.
Measure: Number; unit: percentage of participants with DLT
Arm/Group | Phase I | Phase II
Number analyzed (Participants) | 12 | 0
percentage of participants with DLT
  2.5 mg/day | 0 |
  3.0 mg/day | 0 |
  3.5 mg/day | 66 |

2. Secondary Outcome: Number of Participants With Treatment Related Adverse Events.
Description: Adverse events (AE) that are classified as either possibly, probably, or definitely related to study treatment according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE version 3.0). The maximum grade for each type of AE will be recorded for each patient. The number of participants with grade 3 or higher adverse events at least possibly related to study treatment are reported here.
Time Frame: During treatment and every 6 months until 3 years from registration or progression.
Population: None of the Phase I participants were used for this primary endpoint. All 65 Phase II participants were evaluable for this endpoint.
Measure: Number; unit: participants
Arm/Group | Phase II | Phase I
Number analyzed (Participants) | 65 | 0
participants
  Grade 3 or Higher | 6 |
  Grade 4 or Higher | 3 |
  Grade 5 | 0 |

3. Secondary Outcome: Duration of Response Time
Description: Duration of response is defined as the date at which the patient's objective status is first noted to be a CR, PR or CI to the date progression is documented (if one has occurred) or to the date of last follow-up(for those patients who have not progressed).
Time Frame: Time from response to disease progression, intolerance of study drug, or death.
Population: None of the Phase I participants were evaluable for this endpoint. Sixty-five (65) participants were recruited for the Phase II portion. Results presented here are on the 9 Phase II patients who responded to treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II | Phase I
Number analyzed (Participants) | 9 | 0
Months | 5.6 [1.9 to 13.8] |

4. Secondary Outcome: Time to Response
Description: The time to response is defined as the time from study registration to the first date at which the patient's objective status was classified as a response (CR, PR or CI). In patients who do not achieve a response, time to response will be censored at the patient's last evaluation date. The distribution for each of these event-time variables (duration of response and time to response) will be estimated by Kaplan-Meier curves.
Time Frame: Time from registration to the first date of response within twelve 28-day cycles of treatment.
Population: None of the Phase I participants were evaluable for this endpoint. Sixty-five (65) patients were recruited for the Phase II portion. Only 9 of the 65 patients achieved a response. Thus, the median of time to response and the upper limit of 95% confidence interval are not attainable.
Arm/Group | Phase II | Phase I
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Best Overall Response Over the First 6 Cycles of Treatment
Description: Response evaluation:
  Complete Remission (CR):
  Neutrophil count between 1 to 10 x 10^9/L without peripheral blasts in blood or bone marrow.
  Partial Hematologic Response/Partial Remission (PR):
  Increase in neutrophil by 50% + above 10^9/L for neutropenia)
  Clinical Improvement (CI):
  Increase in Neutrophil count, hemoglobin, platelet count or reduction in blood/marrow blasts.
Time Frame: Every cycle of treatment for 6 cycles. Each cycle is 28 days.
Population: None of the participants from the Phase I cohort were analyzed for this endpoint. All 65 Phase II participants were evaluable for this endpoint and included in the analysis.
Measure: Number; unit: participants
Arm/Group | Phase II | Phase I
Number analyzed (Participants) | 65 | 0
participants
  Complete Remission | 0 |
  Partial Remission | 0 |
  Clinical Improvement | 9 |

ADVERSE EVENTS:
Time Frame: Every 28 day cycle while on treatment (up to 12 cycles).
Description: The primary endpoint for the Phase I cohort of participants was to determine the MTD based on the frequency of DLTs at increasing dose levels. The adverse events in the Phase I cohort were summarized as the Phase I primary endpoint. Here, we report adverse events of all 65 Phase II participants.
Arm/Group | Phase II
Serious Adverse Events (participants affected / at risk) | 19/65
Other Adverse Events (participants affected / at risk) | 65/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II (N=65)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Infectious meningitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Upper respiratory infection (Infections and infestations) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II (N=65)
Hemoglobin decreased (Blood and lymphatic system disorders) | 53 (214)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (19)
Nausea (Gastrointestinal disorders) | 9 (16)
Vomiting (Gastrointestinal disorders) | 3 (4)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 65 (477)
Localized edema (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 15 (54)
Neutrophil count decreased (Investigations) | 27 (196)
Platelet count decreased (Investigations) | 43 (274)
Blood uric acid increased (Metabolism and nutrition disorders) | 7 (11)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 18 (81)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 20 (36)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes